CLINICAL TRIAL: NCT02317159
Title: Efficacy and Safety of Imatinib Mesylate as First-line Treatment for the Patients With Chronic Phase of Chronic Myeloid Leukemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cttq (Industry)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMAGE-201
Record Dates: First submitted 2014-12-11; First posted 2014-12-15 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- imatinib，Capsule (Experimental): 400mg imatinib qd
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — 400mg imatinib qd PO

SUMMARY:
This is a efficacy and safety study of imatinib Mesylate Capsule as First line treatment in patients with chronic phase of Chronic Myeloid Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18；
* The new diagnosis of CML patients in six months；
* No proof of extra-medullary infiltration of leukemia；
* ECOG PS score：0-2；
* Hepatic and renal functions are normal，Serum bilirubin≤1.5*ULN, serum ALT and AST≤2.5*ULN, serum Cr≤1.5*ULN;
* Do not receive the treatment of anti-CML；
* Subjects signed informed consent form in line with GCP requirements。

Exclusion Criteria:

* Pregnant or lactating women；
* Received TKIs any time before；
* Failure to control systemic infection or multiple organ failure；
* According to the investigator's judgment, there are concomitant diseases with a serious safety hazard or affect the patients completed the study；
* Being diagnosed with other malignancies in the prior 12 months；
* Have a history of neurological or psychiatric disorders, including epilepsy or dementia；
* Known or suspected allergy to imatinib；
* BSA≤1.5m2；
* Using other experimental drugs or participating in other clinical trials in the prior one months。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
major molecular response | 2 years
  the rate of major molecular response in two years

SECONDARY OUTCOMES:
complete cytogenetics response | 1 years
  the rate of complete cytogenetics response in one years
over survival | 2 years
  the rate of over survival in two years
progress free survival | 2 years
  the rate of progress free survival in two years